CLINICAL TRIAL: NCT01687543
Title: Probiotics for Reduction of Colonisation With Clostridium Difficile in Antibiotic Treated Intensive Care Patients
Brief Title: Probiotics for Reduction of Infections With Clostridium Difficile in Critically Ill Patients
Acronym: ProbiEnt
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Too low inclusion rate and several sites did not comply
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ProENT11
Record Dates: First submitted 2012-08-28; First posted 2012-09-19 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Clostridium Difficile Colonisation; Impact of Enteral Probiotics on Certain Lab Parameters
Keywords: Clostridium difficile; WBC; CRP; Lactate; Urea; Creatinine
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotics (Experimental): Patients will be given a mixture of maltodextrin ( a starch product often used i alimentary products) and two strains of probiotic bacteria ( L. plantarum 299 and L. plantarum 299v ) dissolved in water through a nasogastric tube. Patients randomized 1:1 between groups
  Interventions: Dietary Supplement: L. plantarum 299 and L. plantarum 299v (+maltodextrin)
- Control (Placebo Comparator): Patients will be given only the dissolved maltodextrin in water through the nasogastric tube. Patients randomized 1:1 between groups
  Interventions: Other: Maltodextrin

INTERVENTIONS:
Dietary Supplement: L. plantarum 299 and L. plantarum 299v (+maltodextrin) — A suspension of Lactobacillus plantarum 299 and Lactobacillus plantarum 299v together with maltodextrin is distributed to the patients twice a day.
  Other Names: Lactobacillus plantarum 299; Lactobacillus plantarum 299v; Maltodextrin
  Arms: Probiotics
Other: Maltodextrin — A suspension of maltodextrin (as placebo control) is distributed to the patients twice a day.
  Arms: Control

SUMMARY:
Symptoms of Clostridium difficile infection is almost always induced as a complication to the use of antibiotics. Most ICU patients are given antibiotics.

Probiotics has the ability to improve conditions in the gut and it has been shown in some smaller studies that overgrowth of C. difficile can be reduced or prevented.

In this study the intention is to show with sufficient statistical power that a mixture of two otherwise well studied probiotic strains reduces or prevents the incidence of emerging colonisation with C. difficile in critical ill patients on antibiotics.

Half of the patients will be given a mixture of Lactobacillus plantarum 299 and Lactobacillus plantarum 299v twice daily and the rest a placebo mixture.

Rectal swabs or faeces will be analysed for C.difficile and its toxins and the incidence of new cases will be compared for the two groups.

White blood cells (WBC´s), C reactive protein (CRP), lactate, urea, and creatinine will be followed daily as well as antibiotics, corticosteroids and all acid reducing medication.

Nutrition, enteral and total, and bowel habits will be recorded.

DETAILED DESCRIPTION:
Infections with Clostridium difficile is considered to be the most frequent health care associated bacterial infection. Almost all cases are connected to the use of antibiotics.

The spectra of symptoms of infection reaches from loose stools to sepsis and death. It is estimated that about 5% of the population are carriers without symptoms.

Elderly people are more likely to be diagnosed with C. difficile infections and as about 50 % of ICU admissions (at least in Sweden) are patients aged 64 years or older C. difficile is also an ICU issue.

Probiotic bacteria given to antibiotic treated patients results in fever cases of infection with C. difficile as we and others have shown in some small studies. Due to a low statistical power in our former study this multicentre study is calculated to be large enough to fulfil statistical requirements.

Adult patients with an expected length of stay in intensive care for three days or more can be included.

Primary objective is to find emerging cases of colonisation with C. difficile and consequent symptoms of infection such as diarrhoea.

Cultures and toxin analyses will be taken at inclusion and every second day till day 13 and then every third or fourth day depending on length of ICU stay. Positive cases will be given antibiotics according to normal routines.

No other cultures are collected per protocol but all cultures will be recorded and results will be analysed in order to find any connection between treatment and reduction of secondary infections.

In our earlier small study we found an improved and normalised gut barrier function for those patients that were given probiotic bacteria compared to a worsened, scattered pattern for the placebo group. This is probably why we found that inflammatory parameters improved for the probiotics group while those parameters remained elevated for the control patients. The same goes for creatinine, urea and lactate. This is why we will record those parameters together with blood gas analyses in this expanded study.

Antibiotics and medication with corticosteroids, proton pump inhibitors or other acid reducing preparations, All nutritive prescriptions (enteral formulas and IV solutions as well as medical preparations containing glucose or fat) will be recorded and compared to actually given nutrients.

Bowel movements frequency and consistency will be recorded and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Anticipated need for intensive care 3 days or longer
* Patients condition allowing enteral nutrition to be started within 24 h from ICU admission
* Antibiotics on-going or planned

Exclusion Criteria:

* Known positive test for Clostridium difficile within the last week
* Known ulcers in the mouth, oropharynx, esophagus and stomach
* Known immune deficiencies
* Enteral nutrition contra indicated
* Pancreatitis as admission diagnosis at the hospital or at the ICU
* ICU admission earlier during this period of illness Patient being moribund

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-06; Primary Completion 2017-06 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Differences in emerging cases of Clostridium difficile | Throughout the ICU stay, expected mean LOS 10 days
  Emerging cases of Clostridium difficile, identified as positive cultures and/or toxin tests

SECONDARY OUTCOMES:
White blood cells | Throughout the ICU , expected mean LOS 10 days
  Samples taken at admission or inclusion and then daily
C Reactive Protein | Throughout the ICU , expected mean LOS 10 days
  Samples taken at admission or inclusion and then daily
Creatinine | Throughout the ICU , expected mean LOS 10 days
  Samples taken at admission or inclusion and then daily
Urea | Throughout the ICU , expected mean LOS 10 days
  Samples taken at admission or inclusion and then daily
Lactate | Throughout the ICU , expected mean LOS 10 days
  Samples taken at admission or inclusion and then daily
Ventilator days | Throughout the ICU stay, expected mean LOS 10 days
  Records are held for how long the patients require mechanical ventilation
Length of stay ICU | Length of ICU stay, about 10 days in accordance with a prior similar study
  Length of stay is recorded for the ICU as well as for the Hospital stay
Length of Hospital stay | Within six months from date of ICU admission
  Length of stay is recorded for the Hospital as well as for the ICU stay
Survival | Six months
  For participating patients the status of survival or non survival at days 28 and 180 (six months) will be recorded
Diarrhea and obstipation | Throughout the ICU stay, expected mean LOS 10 days
  As ICU patients tend to display diarrhea as well as obstipation the frequency and consistency of stools will be recorded.
  Probiotics are anticipated to stabilise bowel function

CONTACTS AND LOCATIONS:
Overall Officials: Bengt Klarin, MD, PhD, Principal Investigator — Lund University, Lund, Sweden
Locations (4):
- Sweden (4):
  - Intensive Care Unit, Helsingborg Hospital, Helsingborg
  - Intensive Care Unit, Kristianstad Central hospital, Kristianstad
  - Lund University Hospital, Lund
  - Dept of Anesthesia & Intensive Care, University Hospital of Norrland, Umeå

REFERENCES:
- [Background] Klarin B, Wullt M, Palmquist I, Molin G, Larsson A, Jeppsson B. Lactobacillus plantarum 299v reduces colonisation of Clostridium difficile in critically ill patients treated with antibiotics. Acta Anaesthesiol Scand. 2008 Sep;52(8):1096-102. doi: 10.1111/j.1399-6576.2008.01748.x. PMID 18840110
- See also: Producers of the study products — http://www.probi.se